CLINICAL TRIAL: NCT02380261
Title: Assessment Of The Skin And Ocular Tolerance Of The Product Systane® Lid Wipes (050343-01) And Assessment Of The Study Subject Acceptance, Under Normal Use Conditions
Brief Title: A Clinical Study of Systane® Lid Wipes in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: NOVARTIS BIOCIENCIAS S/A (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: EXR338-P001
Record Dates: First submitted 2015-02-27; First posted 2015-03-05 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-08

CONDITIONS: Ocular Tolerance; Skin Tolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane (Experimental): Systane® Lid Wipes, 1 per eyelid, used once and discarded after each use, for 21 days
  Interventions: Other: Systane® Lid Wipes

INTERVENTIONS:
Other: Systane® Lid Wipes — Commercially-marketed, individually-packaged, pre-moistened eyelid wipe for daily cleaning

SUMMARY:
The purpose of this study is to verify the skin and ocular tolerance of the product Systane® Lid Wipes.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent.
* Agree to adhere to the procedures and requirements of the study.
* Wears makeup daily.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Ocular conditions as specified in protocol.
* Medical conditions as specified in protocol.
* Skin conditions as specified in protocol.
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alcon Brazil
Locations (1):
- Novartis Biociencias SA, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in Brazil.
Pre-assignment Details: Thirty-five participants were enrolled in this study. This reporting group includes all enrolled participants (35).
Period: Overall Study
Arm/Group | Systane
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Arm/Group | Systane
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  Age 18-70 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Contact-dermatitis Adverse Reaction
Description: Participants were assessed by a dermatologist. Contact-dermatitis adverse reaction was characterized by the presence of one or more of the following symptoms or signs: strong itching sensation, erythema, edema, desquamation, papules or vesicles. Both eyes contributed to the analysis.
Time Frame: Day 21
Population: This analysis population includes all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Systane
Number analyzed (Participants) | 35
participants | 0

2. Primary Outcome: Number of Participants With Ocular Clinical Signs and Discomfort Sensations
Description: Participants were assessed by an ophthalmologist. Ocular clinical signs included palpebral edema, conjunctival edema, orbicular secretion, keratoconus, blepharitis, meibomitis, pterygium, hyperemia, chemosis, keratitis, secretion and lacrimation. Both eyes contributed to the analysis.
Time Frame: Day 21
Population: This analysis population includes all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Systane
Number analyzed (Participants) | 35
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of participation in the study (up to 21 days). This analysis group includes all enrolled participants. Ocular AEs are presented for both study eye and non-study eye combined.
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a product and that does not necessarily have a causal relationship with this treatment. All AEs were obtained as solicited and spontaneous comments from the study participants and through regular investigator assessment throughout the study.
Arm/Group | Systane
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.